CLINICAL TRIAL: NCT05202912
Title: A Randomized, Open-label, Single-dose, Crossover Phase 1 Clinical Trial to Evaluate the Effects of Food or Ethnicity on the Pharmacokinetics and Safety/Tolerability of IDX-1197 After Single Oral Administration in Healthy Male Korean, Chinese, and Caucasian Volunteers
Brief Title: Food Effect Study of IDX-1197 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-VDP-104
Record Dates: First submitted 2021-12-16; First posted 2022-01-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-01

CONDITIONS: Healthy Male
Keywords: 1197; IDX-1197; venadaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A(Food effect) (Other)
  Interventions: Drug: IDX-1197(After a meal)
- Cohort B(Single dose) (Other)
  Interventions: Drug: IDX-1197(fasting)

INTERVENTIONS:
Drug: IDX-1197(After a meal) — randomized, open-label, single-dose, 2-period, 2-sequence crossover study in healthy male Korean and Caucasian volunteers
  Arms: Cohort A(Food effect)
Drug: IDX-1197(fasting) — open-label, single-dose study in Chinese male volunteers
  Arms: Cohort B(Single dose)

SUMMARY:
Study to Evaluate the Effects of Food or Ethnicity on the Pharmacokinetics and Safety/Tolerability of IDX-1197 After Single Oral Administration in Healthy Male Korean, Chinese, and Caucasian Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male Korean, Chinese, or Caucasian adults at the age of ≥19 to ≤50 years old at the time of written informed consent:
2. Body weight ≥55.0 kg AND body mass index (BMS) ≥18.0 kg/m2 to <30.0 kg/m2 at screening: BMI(kg/m2) = body weight (kg) / {height (m)}2
3. The subject must voluntarily decide to participate in the study after being informed of, and fully understanding, details of the study; written informed consent must be obtained prior to any of the screening procedures.
4. Eligible for this study as determined by the investigator based on physical examinations, clinical laboratory tests, and interviews.

Exclusion Criteria:

1. Evidence or history of clinically significant hepatic, renal, neurological, respiratory, endocrine, blood and tumor, cardiovascular, urinary, and psychiatric disorders.
2. Evidence or history of gastrointestinal disorders (gastrointestinal ulcer, gastritis, gastrodynia, gastroesophageal reflux disease, Crohn's disease, etc.) that might affect the safety and PK of IP and/or history of gastrointestinal surgery (except for simple appendectomy and hernia repair).
3. Hypersensitivity to drugs or history of any clinically significant hypersensitivity.
4. Any of the following screening test results:

   * Hemoglobin level < 12.0 g/dL
   * Creatinine clearance: <60 mL/min/1.73m2 as calculated by the equation of Modification of Diet in Renal Disease
   * QTc interval: > 450 ms
   * Positive serum tests (hepatitis B, hepatitis C, human immunodeficiency virus, syphilis)
5. Screening systolic blood pressure <90 mmHg or >150 mmHg and/or diastolic blood pressure <60 mmHg or >100 mmHg as measured in sitting position after ≥3 minutes of rest.
6. History of drug abuse or a positive urine screening test for drugs of abuse.
7. Prior or expected treatment with any prescription drugs or herbal medicine within 2 weeks and/or any over the counter drugs, health functional foods, or vitamins within 1 week prior to the planned first IP dosing (individuals who are determined to be eligible at the discretion of the investigator based on other criteria will be allowed to participate in the study).
8. Treatment with drug metabolizing enzyme inducers and/or suppressors such as barbitals within 1 month prior to the planned first IP dosing.
9. Having participated in another clinical trial or a bioequivalence study and administered any IP within 6 months prior to the planned first IP dosing in the present study.
10. Whole blood donation within 2 months and/or apheresis donation within 1 month and/or blood transfusion within 1 month prior to the planned first IP dosing.
11. Continuous, excessive caffeine intake or continuous alcohol intake or unable to refrain from caffeine/alcohol consumption during hospitalization.
12. Current smoker (individuals who stopped smoking 3 months prior may be included in the study) or unable to stop smoking from 3 months prior to the planned first IP dosing to the last hospital discharge.
13. Having had any foods containing grapefruits from 24 hours prior to hospital admission to discharge in each period/cohort and/or unable to refrain from having foods containing grapefruits during the same period of time.
14. Unable to refrain from having foods containing caffeine (coffee, tea [black tea, green tea, etc.], carbonated drink, coffee milk, nutrients and tonics, etc.) from 24 hours prior to hospital admission to discharge in each period/cohort.
15. Individual or his spouse/partner who is unable to use medically acceptable methods of contraception throughout the study plus for at least 3 months from the last IP dosing and who does not agree not to donate sperm during the same period of time.
16. Ineligible for study participation in the opinion of the investigator for other reasons including clinical laboratory test results.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
Cmax of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured
AUClast of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured

SECONDARY OUTCOMES:
AUCinf of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured
Tmax of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured
t1/2 of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured
CL/F of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured
Vd/F of IDX-1197 | through study completion, an average of 1 year
  PK parameters will be assessed using plasma IDX-1197 concentrations measured

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided